CLINICAL TRIAL: NCT02781116
Title: Risk Assessment Tool for Breast Cancer in Saudi Arabia
Brief Title: Risk Assessment Tool in Saudi Arabia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Guard Health Affairs (Other Government)
Responsible Party: Principal Investigator, Nagham Sheblaq, CCRP, BsC. pharma, Research Supervisor, National Guard Health Affairs
Other Study IDs: Risk Assessment
Record Dates: First submitted 2016-03-31; First posted 2016-05-24 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will have great impact and influence in the medical setting as the targeted model that will be derived from this study will be the pioneer in our region. This model will be beneficial in identifying risk factors and its association with the Arab women population. Furthermore, it will bring chemotherapy prevention once the risk factors and the model are established. Risk factors maybe different from those identified in western women by Gail and IBIS Models

DETAILED DESCRIPTION:
Breast cancer is the most common cancer worldwide. Incidence and mortality have reached a plateau and appear to be dropping in both United States and parts of Western Europe. This decline has been attributed to several factors such as early detection through the use of screening mammography and appropriate use of systemic adjuvant therapy. Breast cancer is a disease and that is predominantly influenced by risk factors which can be allocated to one of four groups: first, family history / genetic which accounts for 15% of all breast cancer cases. The second group which is the most known risk factor for breast cancer can be linked to hazardous effects of hormonal exposures such as early age at menarche, late age at menopause, small number of children and nulliparity, late age at first birth and little or no breast feeding. Long term use of hormone replacement therapy but apparently not long term use of oral contraceptives is also important. The third group is high mammographic breast density which has been shown to be one of the most significant markers of breast cancer risk and the fourth group is having a history proliferative benign breast disease.

Recently, there is a belief that overall caloric intake and obesity in particular with weight gain are related to increased breast cancer risk with different effects between pre and post menopausal women. Also physical activity appears to be important, above and beyond its effect on weight.

There are scattered studies about breast cancer risk factors in the Arab region. One study was published on March 2002 which investigates risk factors associated with breast cancer in Jordanian women while some studies associate diet with breast cancer. The known / well-established risk factors in the Western countries have not bee systematically validated or proven to play a role in Arab women with breast cancer. Therefore, there is no known risk assessment tool that is applicable to our patient population. No model has not been created yet synthesizing the breast cancer risk factors in Arab women.

Research Impact:

This study will have great impact and influence in the medical setting as the targeted model that will be derived from this study will be the pioneer in our region. This model will be beneficial in identifying risk factors and its association with the Arab women population. Furthermore, it will bring chemotherapy prevention once the risk factors and the model are established. Risk factors maybe different from those identified in western women by Gail and IBIS Models

ELIGIBILITY:
Inclusion Criteria:

* All female patients attended the breast cancer screening center

Exclusion Criteria:

* Refusal of participation

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All female patients attended the breast cancer screening center
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
The number of new breast cancer identified with the new risk assessment model that more applicable for our population | 5 years

SECONDARY OUTCOMES:
1. The number of new breast cancer cases using Tyrer Cuzick models that applied in our patients | 5 years
Collect number of IVF and ovarian stimulation in prediction of breast cancer | 5 years
Collect BMI measure in kg/m^2 | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Omalkhair Abulkhair, Principal Investigator — Ministry of National Guard Health Affairs
Locations (1):
- King Abdul Aziz Medical City for National Guard Health Affairs, Riyadh, Saudi Arabia